CLINICAL TRIAL: NCT04518696
Title: Suprachoroidal Buckling for the Management of Rhegmatogenous Retinal Detachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fang Wang (Other)
Responsible Party: Sponsor-Investigator, Fang Wang, Chief of department of ophthalmology, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08.01.10002
Record Dates: First submitted 2020-08-13; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- suprachoroidal buckling treatment group (Experimental): suprachoroidal buckling for therapy of rhegmatogenous retinal detachment
  Interventions: Procedure: suprachoroidal buckling

INTERVENTIONS:
Procedure: suprachoroidal buckling — Location, marking and freezing of the retinal tear on the scleral side . Subretinal fluid is released from the outside of the sclera as needed. In the quadrant of the retinal tear, the spherical conjunctiva was opened and the radial full-thickness scleral incision (3mm)was made about 8-13mm away from the retinal tear. After the choroid was exposed, a "pocket" is formed by injecting some viscoelastic agent into the posterior edge of the sclera and separating the choroid from the sclera using the Healon packaged cannula (No.27 Rycroft cannula). The Healon 5 syringe was connected with a 450-um special tube . The cannula is inserted into the supragromal space under microscopic and was scaned by iOCT . Once confirmed in accord with the needle position, sodium hyaluronate injection, usually need 0.2 mL to 0.5 mL, application of anterior chamber puncture or subretinal fluid stable intraocular pressure. Exit the duct and close the incision with scleral presutures.

SUMMARY:
Study of novel surgical technic-suprachoroidal buckling for therapy of rhegmatogenous retinal detachment.It was excpted to reattached the retina and improve visual function of rhegmatogenous retinal detachment patients.

DETAILED DESCRIPTION:
The operation was performed under a surgical microscope with a 25G Chandelier light source and a wide-field observation system to observe the fundus.Location, marking and freezing of the retinal tear on the scleral side .

Subretinal fluid is released from the outside of the sclera as needed. The spherical conjunctiva was opened and the radial full-thickness scleral incision (3mm)was made about 8-13mm away from the retinal tear. A "pocket" is formed by injecting some viscoelastic agent into the posterior edge of the sclera and separating the choroid from the sclera using the Healon packaged cannula (No.27 Rycroft cannula). The Healon 5 syringe was connected with a 450-um special tube (a 23 caliber curved tube with olive tip). The cannula is inserted into the supragromal space under microscopic and was scaned by iOCT . Monitor the location of retinal tear during intubation in real time, and adjust the position of the needle: posterior margin of the tear. Once confirmed in accord with the needle position, sodium hyaluronate injection, injection needles to in front of shift to injection, until the tear was completely surrounded in viscoelastic agent to create the choroid crest, usually need 0.2 mL to 0.5 mL. Exit the duct and close the incision with scleral presutures.

ELIGIBILITY:
Inclusion Criteria:

* (1) Clinical diagnosis of rhegmatogenous retinal detachment; (2)myopia < 600 degrees； (3) retinal tear were peripheral part, non-proliferative round hole or horseshoe tear, single or multiple tears within one oclock area; (4) PVR grading: Grade A, B, C1, C2; (5) Subretinal fluid was confined around the tear. (6)phakic.

Exclusion Criteria:

* (1)Cataract, corneal degeneration, genetic diseases; (2)History of internal eye surgery; (3)The other eye was blind; (4)Postoperative follow-up could not be scheduled; (5)Systemic diseases (asthma, heart failure, myocardial infarction, liver failure, kidney failure and other serious diseases); (6)History of aspirin and other anticoagulant drugs; (7)Severe adverse reactions and systemic diseases occurred during follow-up.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Retina reattachment | 3 months post operation
  Number of participants who achieved retina reattachment assessed by fundus photography，b-scan ultrasonography and optical coherence tomography.
Best Corrected visual Acuity (BCVA） | 3 months post operation
  Patients' best corrected visual acuity assessed by logarithmic visual acuity charts.
Intraocular pressure (IOP) | 3 months post operation
  Patients' IOP assessed by noncontact tonometer
Treatment-related adverse event | 3 months post operation
  Number of participants with treatment-related adverse events（including suprachoroidal hemorrhage, subretinal hemorrhage, vitreous hemorrhage）

SECONDARY OUTCOMES:
Retina reattachment | 12 months post operation
  Number of participants who achieved retina reattachment assessed by fundus photography，b-scan ultrasonography and optical coherence tomography.
Best Corrected visual Acuity (BCVA） | 12 months post operation
  Patients' best corrected visual acuity assessed by logarithmic visual acuity charts.
Intraocular pressure (IOP) | 12 months post operation
  Patients' IOP assessed by noncontact tonometer
Treatment-related adverse event | 12 months post operation
  Number of participants with treatment-related adverse events（including suprachoroidal hemorrhage, subretinal hemorrhage, vitreous hemorrhage）

CONTACTS AND LOCATIONS:
Overall Officials: Fang Wang, MD,phD, Principal Investigator — Department of ophthalmology, Shanghai Tenth People's Hospital

IPD SHARING:
Plan to Share IPD: Yes
Summarize the experience and deficiency of clinical research process and operation technology, and complete the preliminary report of clinical research.
Supporting Information: Study Protocol, CSR
Time Frame: 2021.01.31 The follow-up work of the study subjects was completed, and statistical analysis was conducted 2021.10.31 Continue to complete the follow-up of all patients, and make statistical analysis of all the data, and scientifically evaluate the results; Summarize the experience and deficiency of clinical research process and operation technology, and complete the preliminary report of clinical research.
Access Criteria: All access

REFERENCES:
- [Background] Antaki F, Dirani A, Ciongoli MR, Steel DHW, Rezende F. Hemorrhagic complications associated with suprachoroidal buckling. Int J Retina Vitreous. 2020 Apr 16;6:10. doi: 10.1186/s40942-020-00211-6. eCollection 2020. PMID 32318273
- [Result] Szurman P, Boden K, Januschowski K. Suprachoroidal Hydrogel Buckling as a Surgical Treatment of Retinal Detachment: Biocompatibility and First Experiences. Retina. 2016 Sep;36(9):1786-90. doi: 10.1097/IAE.0000000000001116. No abstract available. PMID 27429389
- [Result] Mikhail M, El-Rayes EN, Kojima K, Ajlan R, Rezende F. Catheter-guided suprachoroidal buckling of rhegmatogenous retinal detachments secondary to peripheral retinal breaks. Graefes Arch Clin Exp Ophthalmol. 2017 Jan;255(1):17-23. doi: 10.1007/s00417-016-3530-8. Epub 2016 Nov 16. PMID 27853956
- [Result] El Rayes EN, Mikhail M, El Cheweiky H, Elsawah K, Maia A. SUPRACHOROIDAL BUCKLING FOR THE MANAGEMENT OF RHEGMATOGENOUS RETINAL DETACHMENTS SECONDARY TO PERIPHERAL RETINAL BREAKS. Retina. 2017 Apr;37(4):622-629. doi: 10.1097/IAE.0000000000001214. PMID 27482642
- [Result] Boden KT, Januschowski K, Szurman P. [Suprachoroidal Hydrogel Buckle - a New Minimal-Invasive Technique in Treatment of Rhegmatogenous Retinal Detachment]. Klin Monbl Augenheilkd. 2019 Mar;236(3):308-312. doi: 10.1055/s-0043-102947. Epub 2017 Apr 4. German. PMID 28376555